CLINICAL TRIAL: NCT06810661
Title: Managing Frailty Through Mobilization in Males and Female Inpatients with Cardiovascular Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Vitalite Health Network (Unknown)
Responsible Party: Principal Investigator, Myles William O'Brien, Dr., Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 102088 (Event #: 59695)
Record Dates: First submitted 2025-01-27; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Diseases; Frailty
Keywords: Frailty management; mobilization; sex differences; physical activity; cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases; Frailty; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Males (Experimental): A team of Kinesiologists visit the patients daily from admission to discharge to promote movement and help them mobilize to the best of their capabilities (e.g., walking, standing, or sitting on the edge of the bed).
  Interventions: Behavioral: Mobility promotion
- Females (Experimental): A team of Kinesiologists visit the patients daily from admission to discharge to promote movement and help them mobilize to the best of their capabilities (e.g., walking, standing, or sitting on the edge of the bed).
  Interventions: Behavioral: Mobility promotion

INTERVENTIONS:
Behavioral: Mobility promotion — At the Georges-L. Dumont hospital, a patient mobilization program has been introduced on floor 4C that embeds Kinesiologists within care to visit patients daily. A team of Kinesiologists visit the patients daily to promote movement and help them mobilize to the best of their capabilities (e.g., walking, standing, or sitting on the edge of the bed). The investigators propose to continue this individualized model but incorporate activity and frailty measures in males and females with cardiovascular disease.

SUMMARY:
Frailty describes the overall health of a person. Inpatients with cardiovascular problems have a higher risk for frailty - or the sick are more likely to get sicker - causing longer hospital stays, hospital readmission, and death. Females are particularly vulnerable to these problems, generally displaying higher frailty levels than males. In hospital, patients spend almost all their time in bed, and this lack of movement worsens cardiovascular and musculoskeletal health, sometimes lengthening patients' hospital stay and priming them for another cardiovascular event. Prolonged sedentary time may be more detrimental on frailty among females than males. The proposed pilot project will test if an in-hospital General Medicine mobilization program reduces frailty (measure of overall health) in male and female inpatients with cardiovascular disease. A Kinesiologist will provide daily check-ins and promote daily movement (e.g., standing more, resistance bands, physical activity promotion, etc.). The investigators expect both males and females will lower their frailty levels, but given their higher frailty levels in general and because females are typically less active than males, the investigators expect the intervention's effects to be greatest among females. Sixty patients (30 females) will be recruited. Patients with a major heart problem, projected to be in-hospital for at least 3-days, and can independently provide consent. Frailty will be measured using a validated questionnaire. Participants will also be equipped with activity monitors for 24h/d continuous wear to measure amount of time spent stepping, sitting, and lying. Hospital records will be used for length of stay and readmissions. The investigators will compare the outcomes (activity and frailty) between males and females to determine if the intervention impacted each sex differently. This work will guide improved care plans to decrease frailty and improve health outcomes in both male and female patients with heart problems.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted to unit 4C at the Vitalité Health Network
* Patients who have a cardiovascular disease (e.g., heart failure)
* Those who are projected to be in-hospital for at least 3-days
* Patients who are not in a shared room with another study participant
* Patients who are able to independently provide consent or have a caregiver provide consent
* Can communication in French or English

Exclusion Criteria:

-Patients enrolled in other clinical trials or interventions that might confound the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Frailty | At enrollment and at the end of treatment, approximately 2 weeks
  Frailty will be assessed in each participant using the validated Frailty Index used extensively by our group, which calculates frailty as a proportion of health problems present in each person. A trained researcher will help the patient complete the Frailty Index and measure participants' frailty using the Clinical Frailty Scale (scored from 1 [very fit] to 9 [terminally ill]). This scale ensures us a way to obtain a graded frailty score for participants who might be unable to complete the longer questionnaire with assistance.
Physical Activity & Postures | From enrollment through to the end of treatment, approximately 2 weeks
  Movement will be measured using activPAL inclinometers positioned on the patients' torso, thigh, and shin. Monitors will be waterproofed and attached 24-hr/day for at least 3-days using a clear medical dressing. We have safely attached these devices to patients' skin for longer durations (14+ days). Amount of time spent (minutes/day) spent on different activities including physical activity (e.g., steps, physical activity intensity), upright posture, and detailed sedentary postures (e.g., sitting versus lying time) will be determined via validated, custom software that was developed and openly published by the investigator's group.

SECONDARY OUTCOMES:
Hospital Length of Stay | From date of admission to the hospital until the date they will be discharged hospital (at least 3-days)
Hospital Readmissions | Hospital readmissions within 30 days will be quantified by medical records one-month after hospital discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Georges-L.-Dumont University Hospital CentreDr. Georges-L.-Dumont University Hospital Centre, Moncton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Brien MW, Schwartz BD, Shivgulam ME, Daley WS, Frayne RJ, Kimmerly DS. Higher habitual lying time is inversely associated with vagal-related heart rate variability outcomes in younger adults. Appl Physiol Nutr Metab. 2023 Nov 1;48(11):876-881. doi: 10.1139/apnm-2023-0167. Epub 2023 Jul 10. PMID 37429038
- [Background] O'Brien MW, Daley WS, Schwartz BD, Shivgulam ME, Wu Y, Kimmerly DS, Frayne RJ. Characterization of Detailed Sedentary Postures Using a Tri-Monitor ActivPAL Configuration in Free-Living Conditions. Sensors (Basel). 2023 Jan 4;23(2):587. doi: 10.3390/s23020587. PMID 36679384
- [Background] Church S, Rogers E, Rockwood K, Theou O. A scoping review of the Clinical Frailty Scale. BMC Geriatr. 2020 Oct 7;20(1):393. doi: 10.1186/s12877-020-01801-7. PMID 33028215
- [Background] O'Brien MW, Kimmerly DS, Theou O. Impact of age and sex on the relationship between carotid intima-media thickness and frailty level in the Canadian Longitudinal Study of Aging. J Cardiol. 2023 Aug;82(2):140-145. doi: 10.1016/j.jjcc.2023.01.004. Epub 2023 Jan 20. PMID 36682711
- [Background] Kehler DS, Clara I, Hiebert B, Stammers AN, Hay JL, Schultz A, Arora RC, Tangri N, Duhamel TA. Sex-differences in relation to the association between patterns of physical activity and sedentary behavior with frailty. Arch Gerontol Geriatr. 2020 Mar-Apr;87:103972. doi: 10.1016/j.archger.2019.103972. Epub 2019 Nov 7. PMID 31739110
- [Background] McCarthy C, Warne JP. Gender differences in physical activity status and knowledge of Irish University staff and students. Sport Sci Health. 2022;18:1283-91
- [Background] Humphries KH, Izadnegahdar M, Sedlak T, Saw J, Johnston N, Schenck-Gustafsson K, Shah RU, Regitz-Zagrosek V, Grewal J, Vaccarino V, Wei J, Bairey Merz CN. Sex differences in cardiovascular disease - Impact on care and outcomes. Front Neuroendocrinol. 2017 Jul;46:46-70. doi: 10.1016/j.yfrne.2017.04.001. Epub 2017 Apr 18. No abstract available. PMID 28428055
- [Background] Perez-Zepeda MU, Martinez-Velilla N, Kehler DS, Izquierdo M, Rockwood K, Theou O. The impact of an exercise intervention on frailty levels in hospitalised older adults: secondary analysis of a randomised controlled trial. Age Ageing. 2022 Feb 2;51(2):afac028. doi: 10.1093/ageing/afac028. PMID 35180287
- [Background] Theou O, O'Brien MW, Godin J, Blanchard C, Cahill L, Hajizadeh M, Hartley P, Jarrett P, Kehler DS, Romero-Ortuno R, Visvanathan R, Rockwood K. Interrupting bedtime to reverse frailty levels in acute care: a study protocol for the Breaking Bad Rest randomized controlled trial. BMC Geriatr. 2023 Aug 10;23(1):482. doi: 10.1186/s12877-023-04172-x. PMID 37563553
- [Background] Theou O, Kehler DS, Godin J, Mallery K, MacLean MA, Rockwood K. Upright time during hospitalization for older inpatients: A prospective cohort study. Exp Gerontol. 2019 Oct 15;126:110681. doi: 10.1016/j.exger.2019.110681. Epub 2019 Aug 2. PMID 31382011
- [Background] Romero-Ortuno R, Wallis S, Biram R, Keevil V. Clinical frailty adds to acute illness severity in predicting mortality in hospitalized older adults: An observational study. Eur J Intern Med. 2016 Nov;35:24-34. doi: 10.1016/j.ejim.2016.08.033. Epub 2016 Sep 2. PMID 27596721
- [Background] Vitale C, Jankowska E, Hill L, Piepoli M, Doehner W, Anker SD, Lainscak M, Jaarsma T, Ponikowski P, Rosano GMC, Seferovic P, Coats AJ. Heart Failure Association/European Society of Cardiology position paper on frailty in patients with heart failure. Eur J Heart Fail. 2019 Nov;21(11):1299-1305. doi: 10.1002/ejhf.1611. Epub 2019 Oct 23. PMID 31646718
- [Background] Denfeld QE, Jha SR, Fung E, Jaarsma T, Maurer MS, Reeves GR, Afilalo J, Beerli N, Bellumkonda L, De Geest S, Gorodeski EZ, Joyce E, Kobashigawa J, Mauthner O, McDonagh J, Uchmanowicz I, Dickson VV, Lindenfeld J, Macdonald P. Assessing and managing frailty in advanced heart failure: An International Society for Heart and Lung Transplantation consensus statement. J Heart Lung Transplant. 2023 Nov 29:S1053-2498(23)02028-4. doi: 10.1016/j.healun.2023.09.013. Online ahead of print. PMID 38099896
- [Background] Tanuseputro P, Manuel DG, Leung M, Nguyen K, Johansen H; Canadian Cardiovascular Outcomes Research Team. Risk factors for cardiovascular disease in Canada. Can J Cardiol. 2003 Oct;19(11):1249-59. PMID 14571310
- [Background] Afilalo J, Karunananthan S, Eisenberg MJ, Alexander KP, Bergman H. Role of frailty in patients with cardiovascular disease. Am J Cardiol. 2009 Jun 1;103(11):1616-21. doi: 10.1016/j.amjcard.2009.01.375. Epub 2009 Apr 8. PMID 19463525